CLINICAL TRIAL: NCT01136018
Title: A Prospective Evaluation of Iodinated Contrast Flow Patterns in Caudal Epidurography With Intentional Lateral Caudal Approach
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Kyoung-bong Yoon, Anesthesiology in Severance hospital
Other Study IDs: 4-2010-0016
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Patient Who Needs Epidural Block

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- intentional lateral caudal approach
  Interventions: Procedure: insertion needle via intentionally lateral direction.

INTERVENTIONS:
Procedure: insertion needle via intentionally lateral direction. — evaluation of iodinated contrast flow patterns in caudal epidurography with intentional lateral caudal approach

SUMMARY:
Caudal epidural block is useful not only for regional anesthesia of low abdominal, perineal area or lower extremities but for relieving acute or chronic pain of low back and lower extremities. Recently, there were some reports that there was a difference of the contrast flow pattern during lumbar epidural block according to a location of needle tip in the lumbar epidural space. Therefore, the investigators hypothesize that there is a difference of contrast flow pattern in caudal epidurography when a needle is inserted with intentionally lateral direction.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral radiculopathy

Exclusion Criteria:

* patients with sepsis
* chronic infection
* coagulopathy
* local infection near the sacral hiatus
* the allergy of the contrast
* history of spine surgery, scoliosis and kyphosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
A prospective evaluation of iodinated contrast flow patterns in caudal epidurography with intentional lateral caudal approach | during 10 seconds after obtaining the caudal epidurogram
  Caudal epidural block is useful not only for regional anesthesia of low abdominal, perineal area or lower extremities but for relieving acute or chronic pain of low back and lower extremities. Recently, there were some reports that there was a difference of the contrast flow pattern during lumbar epidural block according to a location of needle tip in the lumbar epidural space. Therefore, the investigator hypothesizes that there is a difference of contrast flow pattern in caudal epidurography when a needle is inserted with intentionally lateral direction.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea